CLINICAL TRIAL: NCT02573519
Title: Gastrointestinal Motility Among Diabetes Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Renewal of PET/CT scanners and slow recruitment
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry); Svend Faelding Humanitarian Foundation (Unknown); Copenhagen University Foundation for Medical Students (Unknown); Hoejmosegaard Foundation (Unknown); Holger Rabitz og Hustru Doris Mary foedt Phillipps Mindelegat (Unknown); Lundbeck Foundation (Other); Wilhelm Frank og Angelina Franks Mindelegat (Unknown); Torben og Alice Frimodts Fond (Unknown); Fonden til Lægevidenskabens Fremme, A.P. Møller Fonden (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1-10-72-54-15
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Autonomic Neuropathy; Gastrointestinal Motility Disorder; Diabetes Mellitus; Change of Transit or Circulation
Keywords: 11C Donepezil PET/CT scan; 3D-Transit; Diabetes Mellitus; Gastrointestinal motility disorder; Diabetic autonomic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — Pyridostigmine Bromide; Cyclin-Dependent Kinase Inhibitor p15

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic patient (Active Comparator): The study consists of four different parts:
  1. 11C Donepezil PET/CT scan
  2. 3D-Transit
  3. 3D-Transit during treatment with pyridostigmine
  4. 3D-Transit after Malone appendicostomy (only diabetic patients who had a Malone-surgery for severe obstipation ordered during standard clinical practice)
  Interventions: Radiation: 11C Donepezil PET/CT scan; Device: 3D-Transit; Drug: 3D-Transit during treatment with Pyridostigmine; Device: 3D-Transit after Malone appendicostomy
- Healthy subjects (Active Comparator): The study consists of two different parts:
  1. 11C Donepezil PET/CT scan
  2. 3D-Transit
  Interventions: Radiation: 11C Donepezil PET/CT scan; Device: 3D-Transit

INTERVENTIONS:
Radiation: 11C Donepezil PET/CT scan — Donepezil binds with high affinity to acetylcholine esterase in the cholinergic synapses. The quantity of density of acetylcholine esterase in the abdominal organs including the intestinal wall are demonstrated by 11C Donepezil PET/CT scan. The PET-signal are measured as Standard-uptake values (SUV) in the internal organs. After 6 hours of fast CT- and PET-scans are performed after injection of iv. contrast and about 500MBq (megabecquerel) [11C]donepezil. The CT scan is used for anatomical location of the internal organs. The scan-field includes the heart and the abdominal organs. Total scan time is about 60 minutes.
Device: 3D-Transit — 3D-Transit: 3D-Transit for minimal invasive and ambulant describing of regional transit times and contractions pattern of the bowel. The motility and the passage time is measured by 3D-Transit The description of location and rotation of the capsule is dynamic and very precise. It permits precise detailed description of the gastrointestinal contraction pattern and regional passage time. 3D-transit consist of three different parts:
  1. A wireless electromagnetic capsule to be swallowed by the subject
  2. A portable detector plate comprising four sensors worn in a belt around the waist
  3. Specific software for visualizing and analyzing data
  Other Names: MTS-2
Drug: 3D-Transit during treatment with Pyridostigmine — 3D-Transit and Pyridostigmine: The motility and the passage time is measured by 3D-Transit (as mentioned above) in diabetic patients during administration of Pyridostigmine 60 mg administrated 4 times with 4 hours between each administration. Pyridostigmine is increasing the amount of cholinergic neurotransmitter and is suggested to have a reversible effect on the cholinergic denervation. The mechanism of action of Pyridostigmine in the human body is well-known and the drug is used as a tool to determine if the disturbance in the guts are reversible in diabetic patients.
  Other Names: MTS-2 with treatment of acetylcholine esterase inhibitor
  Arms: Diabetic patient
Device: 3D-Transit after Malone appendicostomy — 3D-Transit (as earlier described) is performed after Malone appendicostomy. The patients are suppose use the antegrade edema technic during the 3D-transit examination.
  Other Names: MTS-2
  Arms: Diabetic patient

SUMMARY:
Gastrointestinal (GI) symptoms including vomiting, nausea, abdominal pain, constipation or chronic diarrhea affect a large number of patients with diabetes mellitus (DM). Furthermore, abnormal GI transit times restrict correct dosing of medication. Two new methods, in combination only available at Aarhus University Hospital (AUH), allow examination of human whole-gut function with a high degree of detail:

PET-scans (positron emission tomography scans) of cholinergic signaling in the bowel wall The most important nerve fibers stimulating GI peristalsis use acetylcholine as neurotransmitter. The novel PET technique, [11C] Donepezil PET/CT (Donepezil PET/CT scan based on a carbon isotope), developed at AUH, allows in vivo quantification of cholinergic cells within the bowel wall.

3D-Transit With 3D-Transit electromagnetic capsules are followed during their passage through the GI tract. The novel method provides highly detailed information about regional and whole-gut passage times and contractility patterns.

Study protocol 20 healthy subjects and 25 diabetic patients with severe GI symptoms will be included.

1. With [11C]donepezil PET/CT, we aim to describe the degree of cholinergic denervation of the intestine in DM patients with GI severe symptoms.
2. Using 3D-Transit in DM patients before and during intervention with acetyl cholinesterase inhibitor we aim to determine how cholinergic denervation of the intestine contributes to abnormal GI transit patterns.
3. Comparing the transit times of DM patients with either vomiting or diarrhea as main symptoms, we aim to provide pilot data on phenotypes of diabetic GI dysfunction.
4. We aim to explore various aspects of "pan-enteric" dysfunction in DM, including prolonged gastric emptying secondary to severe constipation and delayed small intestinal transit in patients with symptoms of gastroparesis with or without delayed gastric emptying

Perspectives Detailed information about cholinergic denervation in DM and objective classification of the pathophysiology of diabetic GI dysfunction may allow targeted future treatment of individual patients.

DETAILED DESCRIPTION:
Background GI symptoms are extremely common in patients with DM, often with severe consequences for daily activities, ability to work and quality of life. Moreover, GI-dysfunction causes unpredictable absorption of food and oral medication thus making blood-glucose difficult to control and oral medication less effective. Despite of this fact, the pathophysiology of diabetic bowel dysfunction is only scantily described. Rational treatment of GI motility disorders requires detailed knowledge of the underlying mechanisms and the importance of whole-gut evaluation of patients with motility disorders is increasingly recognized.

Contractions of the GI tract are primary stimulated by cholinergic parasympathetic nerves (from the vagus nerve and the sacral nerves) or cholinergic nerves in the enteric nerve system located between the muscle layers in the bowel wall. It is likely that cholinergic denervation is a major factor behind the development of GI dysfunction in DM.

Through collaboration between basic physiologist and clinical researchers we are in the unique international position of having two highly advanced methods for description of GI innervation and motility:

A. [11C]donepezil (Donepezil connected with a carbon isotope) PET tracer to quantify the density of acetylcholine esterase in abdominal organs, including the intestinal wall. The method constitutes the first-ever validated scan-method for in vivo measuring cholinergic denervation of the GI tract.

B. 3D-Transit for minimal invasive and ambulant describing of regional transit times and contractions pattern of the bowel.

Through studies based on the two methods we aim to test the following hypotheses:

1. The [11C]donepezil PET signal of the intestinal wall is weaker than normal in patients with DM and GI symptoms.
2. Compared to healthy controls, patients with diabetes has prolonged transit time through the stomach, the small intestine and the colorectum.
3. Prolonged transit times through the stomach, small intestine and colorectum of diabetic patients are, at least in part, reversible and approach normal during acetylcholine esterase inhibitor treatment.

5. Gastrointestinal dysfunction in DM is "pan-enteric" and assessment of one region is insufficient as clinical evaluation.

Diabetes and dysmotility of the gastrointestinal tract Autonomic neuropathy can affect all parts of the GI tract, which makes specific diagnosis and correct therapy difficult. Diabetes is strongly associated with nausea, vomiting, diarrhea, abdominal pain, constipation and fecal incontinence. The best-investigated aspect of diabetic dysmotility is gastroparesis. It has been reported that one third of patients with DM having delayed emptying of the stomach. However, gastroparesis is usually detected after at least 10 years of diabetes.

The pathophysiology of diabetic gastroparesis is still incompletely described but includes lack of co-coordinated contractions of the stomach, deficient relaxation of the pylorus and fundus of the stomach relaxation. Furthermore both peripheral and central sensory function is abnormal. Small intestine dysfunction in DM is very scantily investigated. Thus, it is still unknown whether patients with diabetic neuropathy primary have rapid or slow passage time through the small intestine. This is important because treatment of the two conditions is opposite.

Autonomic and enteric neuropathy in diabetes The neural control of GI motility is complex. The most essential components are the enteric nervous system located in the bowel wall and parasympathetic nerve fibers from vagus nerve or the sacral nerves. In both systems acetylcholine is the most important stimulating neurotransmitter. It is well known that DM may cause autonomic neuropathy affecting the visceral organs.

Earlier studies of patients with DM have found demyelination, axonal damage and reduced number of motor fibers in vagal nerves. However, the correlation between GI symptoms and other evidences of autonomic neuropathy is poor. Other studies report degeneration of nerve fibers within the enteric nervous system including the Cajal cells (the pacemaker cell of the bowel). Today, it is assumed that diabetic GI dysfunction is caused by a combination of autonomic neuropathy, enteric neuropathy, dysfunction of the Cajal cells, reduced contractility of the intestinal smooth muscle cells and abnormally high blood glucose. The clinical effect of each component is unknown.

Methodological limitations of previous studies of GI dysfunction in diabetes Previous studies, mentioned above, are all observational in design and the changes in nerve or muscle cell function were not correlated to the specific changes in bowel function. Therefore, it has not been possible evaluate the functional effects of neuropathy of specific groups of neurons or lack of specific neurotransmitters. This important aspect will be addressed in the present study.

Most neurons controlling GI motility are located in myenteric plexus deeply in the bowel wall, not available for ordinary biopsies. Thus, most studies of diabetic GI neuropathy have been based on animal models and results cannot directly be applied to humans. Studies of GI contractions and motility patterns under near normal conditions have been difficult to perform because subjects had to be confined to hospital or have catheters inserted. Especially, the small intestine is difficult to access.

[11C]donepezil PET/CT Donepezil binds with high affinity to acetylcholine esterase in the cholinergic synapses.

Parkinson is a disease characterized by noticeable loss of parasympathetic nerve fibers. Like with DM, Parkinson patients often suffer from severe gastroparesis and constipation. We have recently validated [11C]donepezil PET/CT as a measure of the density of acetylcholine esterase in peripheral organs. A high [11C]donepezil PET signal is seen in heart, liver, and pancreas while and medium signal is seen in in the small intestine, and a weak signal in the colon. The intensity of the signal is correlated to areas with known high density of vagal innervation area. In a study of 12 patients with Parkinson´s disease and 12 healthy the patients had a dramatic loss of signal in the small intestine but also a measurable loss in the pancreas. Thus, [11C]donepezil PET constitutes the first validated scan-method for demonstrating parasympathetic denervation in vivo.

Subjects and methods We aim to include 20 healthy subjects and 25 patients with DM and severe GI symptoms (nausea, vomiting, abdominal discomfort, diarrhea or constipation). Standard assessment will be performed prior to inclusion as part of daily clinical practice. Persons with a history of disease within the central nervous system or the gastrointestinal tract and those with a history of major abdominal surgery are excluded.

1. All Subjects will be examined with [11C]donepezil PET/CT to compare the total cholinergic innervation of the gut in patients with DM and healthy.
2. All subjects will be examined with 3D-Transit to compare gastric emptying time, small intestinal transit time, and colorectal transit time in patients with DM and healthy controls.
3. Patients with DM will be examined with 3D-Transit time a second time after administration of the acetylcholine esterase inhibitor Mestinon (60 mg x 4) to determine whether abnormal transit times and patterns are reversible and thus caused by cholinergic denervation.
4. A minority of patients with severe intractable constipation will on clinical indications have a Malone appendicostomy. This procedure ensures efficient emptying of the colon and rectum. These patients will undergo a third examination with 3D-Transit. Comparing this investigation to their first will provide pilot data on to what degree gastroparesis is secondary to severe constipation Health Ethics Committee for Region Middle, Denmark, has approved the project. The protocol has been submitted to "The Danish Health and Medicines Authority".

PET/CT with [11C]donepezil The total radiation dose for the PET/CT is about 7-8 millisievert (mSv), which corresponds to about 2.5 years of background irradiation, or half that of an ordinary diagnostic CT-scan. This radiation dose is linked to a theoretical increased risk for cancer estimated to about 0.05%.

3D-Transit Every capsule (8x21 mm) Capsules emits a electromagnetic field, which is converted to the coordinates (x;y;z;Φ;θ). The coordinates x;y;z defines the distance with few millimeters precision. Φ;θ defines the angle of the magnet in relation to the sensors. The description of location and rotation of the capsule is dynamic and very precise and permits detailed description of the GI-contraction patterns and regional passage time. Artifacts from breathing and physical activity are recorded from a belt around thorax and an accelerometer in the detector. The 3D-Transit method is without discomfort and has only a negligible risk of capsule retention. The investigation is ambulatory and under circumstances close to the subject's everyday life. This is a considerable advantage compared to traditional investigation methods as scintigraphy and manometry. Validity, safety and reproducibility data from 3D-Transit have been published from our group.

The study consists of four different parts. The DM patients examined in 1-3 and few DM patients are able to participate in part 4. The healthy subjects are only examined in the first two parts (1 and 2).

1. 11C Donepezil PET/CT scan
2. 3D-Transit, capsule 1
3. 3D-Transit capsule 2 while taking acetylcholine esterase inhibitor (Pyridostigmine 60 mg four times with 4 hours between each administration.)
4. 3D-Transit capsule 3 after Malone antegrade continence enema

Each part of the study is completed before the next step begins. The study participants are fasting before each study element. DM patients are taking the morning insulin and closely monitored to reach blood glucoses between 4-10 mmol/L

The practical feasibility of the study The Department of Endocrinology at Aarhus University Hospital has specific interest in diabetic neuropathy and patients will be classified according to international standards.

The Department of Hepatology and Gastroenterology, Aarhus University Hospital has a special interest in neurogastroenterology and has established a professorship in this field. The department has close collaboration with the manufacturer of 3D-Transit (Motilis Medica SA, Lausanne, Switzerland) and the research group in London. Through this ongoing collaboration we have been among the pioneers in the development of magnet tracking for description of GI motility.

The PET Center at Aarhus University Hospital is an internationally recognized research unit in this field. The relevant resources are available, including PET/CT scanners, radiochemical facilities for tracer production, software, and computer scientist assistance for analyzing PET-data.

Future perspectives

1. Decreased cholinergic PET signal in the bowel wall of patients suffering from diabetes and severe GI symptoms, in combination with mechanistic data identifying cholinergic neuropathy as a main cause of abnormal transit patterns will have significant international interest and improve future attempts to develop targeted future treatment.
2. Identification of specific phenotypes of diabetic bowel dysfunction will form the basis of larger descriptive studies to allow future stratified treatment.

ELIGIBILITY:
Inclusion Criteria: (only patients)

* Subject is suffering from diabetes
* Gastrointestinal symptoms including diarrhoea, nausea, vomiting, bloating and abdominal discomfort)
* Subject > 18 years of age who possess capacity to understand subject information sheet and give informed consent for participation
* Fasted since midnight until morning 8 o´clock

Exclusion Criteria:

* Dysregulated metabolic disease
* Structuring bowel disease or obvious stenotic symptoms or perforation
* Subject has known swallowing disorders
* Subject has cancer or other life threatening diseases or conditions
* Subject is pregnant or breastfeeding
* Subject has undergone extensive abdominal surgery
* Subject has a abdominal diameter > 140 cm
* Drug abuse or alcoholism
* Bacterial overgrowth
* Subject has known severe cardiovascular or pulmonary diseases (including artificial pacemaker and/or implantable cardioverter-defibrillator (ICD))
* Central nerve system (CNS) surgery
* Patient have infusion pump or other implantable medical device
* Medication (not possible for pausing for 48 hours) or any other disease affecting motility or/and gastroparesis.
* Subjects having MRI within the next four weeks
* Taking corticosteroids during the last month
* Allergic reaction to Pyridostigmine and/or intravenously administrated contrast
* Severe upper gastrointestinal pathology seen by endoscopy
* Blood glucose below 4 mmol/L or higher than 10 mmol/L right before examination
* Bile acid malabsorption or malabsorption in general
* Obstruction of the urinary system
* Severe renal insufficiency (eGFR < 45)
* Peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Difference in Donepezil standard-uptake values (SUV) for the small intestine between diabetic patients and healthy subjects. | Through study completion, an average of 1 year
  The PET signal is measured as standard-uptake values (SUV) in the internal organs. This simple value has earlier been validated as equivalent to more advanced PET kinetic parameters, were an arterial-needle is required. From the CT-scan volume-of-interests of the relevant organs are applied (bowel segments, heart, pancreas) and the SUV-values draw from the PET-scans. SUV in the small intestine are compared between healthy subjects and diabetic patients. SUV is a measure of in vivo quantification of cholinergic cells in the small bowel.
Difference in total gastrointestinal transit time between diabetic patients and healthy subjects | Through study completion, an average of 1 year
  The following parameters are analyzed: Total gastrointestinal transit time (capsule number 1).
  Data from capsule 1 in healthy subjects and diabetic patients will be used for: Comparison of total GI transit times and transit patterns in healthy individuals and diabetic patients.

SECONDARY OUTCOMES:
Measurement of gastric amplitudes | Through study completion, an average of 1 year
  If new software for analysis permits more detailed data analysis. Amplitudes of gastric contractions during awake and sleep will be analyzed.
Measurement of fast movements in the small intestine | Through study completion, an average of 1 year
  If new software for analysis permits more detailed data analysis. Number of "fast movements" in the small intestine will be analyzed.
Measurement of mass movements in colorectum | Through study completion, an average of 1 year
  If new software for analysis permits more detailed data analysis. Number and distance covered by "mass-movements" in colorectum will be analyzed.
Difference in total gastrointestinal transit times in diabetic patients´s 3D-transit with and without Pyridostigmine | Through study completion, an average of 1 year
  3D-Transit data from capsule 1 and 2 (only the diabetic patients): By comparing total GI transit times with and without administration of acetylcholine esterase inhibitor mechanistic data will be obtained to determine if neuropathy of acetylcholine containing neurons is the cause of physiological changes in GI transit times. The primary end-point is difference in total gastrointestinal passage time.
Difference in regional intestinal transit times between diabetic patients and healthy subjects | Through study completion, an average of 1 year
  The following parameters are analyzed: Gastric emptying, small intestinal and colorectal transit time (capsule number 1).
  Data from capsule 1 in healthy and patients will be used for: Comparison of regional GI transit times and transit patterns in healthy individuals and diabetic patients.
Difference in regional transit times in diabetic patients´s 3D-transit with and without Pyridostigmine | Through study completion, an average of 1 year
  The following parameters are analyzed: Gastric emptying, small intestinal and colorectal transit time (capsule number 1 and 2, only in diabetic patients).
  Data from capsule 1 and 2 will be used for: Comparison of regional GI transit times and transit patterns in diabetic patients with and without Pyridostigmine
Difference in regional transit times in diabetic patients´s 3D-transit before and after Malone antegrade continence enema | Through study completion, an average of 1 year
  The following parameters are analyzed: Gastric emptying, small intestinal and colorectal transit time (capsule number 1 and 3, only in diabetic patients with Malone Surgery).
  Data from capsule 1 and 3 will be used for: Comparison of regional GI transit times and transit patterns in diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, Professor, Principal Investigator — Department of Hepatology and Gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SS, Camilleri M, Hasler WL, Maurer AH, Parkman HP, Saad R, Scott MS, Simren M, Soffer E, Szarka L. Evaluation of gastrointestinal transit in clinical practice: position paper of the American and European Neurogastroenterology and Motility Societies. Neurogastroenterol Motil. 2011 Jan;23(1):8-23. doi: 10.1111/j.1365-2982.2010.01612.x. PMID 21138500
- [Background] Bytzer P, Talley NJ, Leemon M, Young LJ, Jones MP, Horowitz M. Prevalence of gastrointestinal symptoms associated with diabetes mellitus: a population-based survey of 15,000 adults. Arch Intern Med. 2001 Sep 10;161(16):1989-96. doi: 10.1001/archinte.161.16.1989. PMID 11525701
- [Background] Maleki D, Locke GR 3rd, Camilleri M, Zinsmeister AR, Yawn BP, Leibson C, Melton LJ 3rd. Gastrointestinal tract symptoms among persons with diabetes mellitus in the community. Arch Intern Med. 2000 Oct 9;160(18):2808-16. doi: 10.1001/archinte.160.18.2808. PMID 11025791
- [Background] Vanormelingen C, Tack J, Andrews CN. Diabetic gastroparesis. Br Med Bull. 2013;105:213-30. doi: 10.1093/bmb/ldt003. Epub 2013 Jan 29. PMID 23363458
- [Background] Jones KL, Russo A, Stevens JE, Wishart JM, Berry MK, Horowitz M. Predictors of delayed gastric emptying in diabetes. Diabetes Care. 2001 Jul;24(7):1264-9. doi: 10.2337/diacare.24.7.1264. PMID 11423513
- [Background] Sarosiek I, Selover KH, Katz LA, Semler JR, Wilding GE, Lackner JM, Sitrin MD, Kuo B, Chey WD, Hasler WL, Koch KL, Parkman HP, Sarosiek J, McCallum RW. The assessment of regional gut transit times in healthy controls and patients with gastroparesis using wireless motility technology. Aliment Pharmacol Ther. 2010 Jan 15;31(2):313-22. doi: 10.1111/j.1365-2036.2009.04162.x. Epub 2009 Oct 8. PMID 19814743
- [Background] Kloetzer L, Chey WD, McCallum RW, Koch KL, Wo JM, Sitrin M, Katz LA, Lackner JM, Parkman HP, Wilding GE, Semler JR, Hasler WL, Kuo B. Motility of the antroduodenum in healthy and gastroparetics characterized by wireless motility capsule. Neurogastroenterol Motil. 2010 May;22(5):527-33, e117. doi: 10.1111/j.1365-2982.2010.01468.x. Epub 2010 Jan 29. PMID 20122128
- [Background] Olausson EA, Brock C, Drewes AM, Grundin H, Isaksson M, Stotzer P, Abrahamsson H, Attvall S, Simren M. Measurement of gastric emptying by radiopaque markers in patients with diabetes: correlation with scintigraphy and upper gastrointestinal symptoms. Neurogastroenterol Motil. 2013 Mar;25(3):e224-32. doi: 10.1111/nmo.12075. Epub 2013 Jan 15. PMID 23316944
- [Background] Rosa-e-Silva L, Troncon LE, Oliveira RB, Foss MC, Braga FJ, Gallo Junior L. Rapid distal small bowel transit associated with sympathetic denervation in type I diabetes mellitus. Gut. 1996 Nov;39(5):748-56. doi: 10.1136/gut.39.5.748. PMID 9014777
- [Background] Sellin JH, Hart R. Glucose malabsorption associated with rapid intestinal transit. Am J Gastroenterol. 1992 May;87(5):584-9. PMID 1595644
- [Background] Guy RJ, Dawson JL, Garrett JR, Laws JW, Thomas PK, Sharma AK, Watkins PJ. Diabetic gastroparesis from autonomic neuropathy: surgical considerations and changes in vagus nerve morphology. J Neurol Neurosurg Psychiatry. 1984 Jul;47(7):686-91. doi: 10.1136/jnnp.47.7.686. PMID 6747645
- [Background] Guo C, Quobatari A, Shangguan Y, Hong S, Wiley JW. Diabetic autonomic neuropathy: evidence for apoptosis in situ in the rat. Neurogastroenterol Motil. 2004 Jun;16(3):335-45. doi: 10.1111/j.1365-2982.2004.00524.x. PMID 15198656
- [Background] Tay SS, Wong WC. Short- and long-term effects of streptozotocin-induced diabetes on the dorsal motor nucleus of the vagus nerve in the rat. Acta Anat (Basel). 1994;150(4):274-81. doi: 10.1159/000147630. PMID 7839795
- [Background] Clouse RE, Lustman PJ. Gastrointestinal symptoms in diabetic patients: lack of association with neuropathy. Am J Gastroenterol. 1989 Aug;84(8):868-72. PMID 2756978
- [Background] Horvath VJ, Vittal H, Lorincz A, Chen H, Almeida-Porada G, Redelman D, Ordog T. Reduced stem cell factor links smooth myopathy and loss of interstitial cells of cajal in murine diabetic gastroparesis. Gastroenterology. 2006 Mar;130(3):759-70. doi: 10.1053/j.gastro.2005.12.027. PMID 16530517
- [Background] Punkkinen J, Farkkila M, Matzke S, Korppi-Tommola T, Sane T, Piirila P, Koskenpato J. Upper abdominal symptoms in patients with Type 1 diabetes: unrelated to impairment in gastric emptying caused by autonomic neuropathy. Diabet Med. 2008 May;25(5):570-7. doi: 10.1111/j.1464-5491.2008.02428.x. PMID 18445170
- [Background] Hopkins DA, Bieger D, deVente J, Steinbusch WM. Vagal efferent projections: viscerotopy, neurochemistry and effects of vagotomy. Prog Brain Res. 1996;107:79-96. doi: 10.1016/s0079-6123(08)61859-2. No abstract available. PMID 8782514
- [Background] Haase AM, Gregersen T, Schlageter V, Scott MS, Demierre M, Kucera P, Dahlerup JF, Krogh K. Pilot study trialling a new ambulatory method for the clinical assessment of regional gastrointestinal transit using multiple electromagnetic capsules. Neurogastroenterol Motil. 2014 Dec;26(12):1783-91. doi: 10.1111/nmo.12461. Epub 2014 Oct 27. PMID 25348504
- [Background] Fynne L, Worsoe J, Gregersen T, Schlageter V, Laurberg S, Krogh K. Gastric and small intestinal dysfunction in spinal cord injury patients. Acta Neurol Scand. 2012 Feb;125(2):123-8. doi: 10.1111/j.1600-0404.2011.01508.x. Epub 2011 Mar 24. PMID 21428967